CLINICAL TRIAL: NCT05556759
Title: Anterior Iliopsoas Muscle Space Block Versus Supra-Iliac Anterior Quadratus Lumborum Block for Analgesia in Total Hip Arthroplasty: A Randomized Controlled Trial
Brief Title: Anterior Iliopsoas Muscle Space Block Versus Supra-iliac Anterior Quadratus Lumborum Block in Total Hip Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Shereen Elsayed Abd Ellatif, associate professor of anesthesia and surgical intensive care, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 9721-18-9-2022
Record Dates: First submitted 2022-09-20; First posted 2022-09-27 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Hip Arthropathy
Keywords: Anterior iliopsoas muscle space block; suprailiac anterior quadratus lumborum block; analgesia; hip arthroplasty
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: The patients will be divided randomly by a computer-generated randomization table into three groups:
  Group C :(Control group) patients will be operated on under general anesthesia. Group IPS: patients will receive anterior IPS block with 30 ml of bupivacaine 0.25% followed by general anesthesia.
  Group Supra-iliac QL: patients will receive supra-iliac anterior QL block with 30 ml of bupivacaine 0.25% followed by general anesthesia.
Who Masked: Participant, Outcomes Assessor
Masking Description: double-blinded(participants and outcome assessors)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Placebo Comparator): patients will be operated on under general anesthesia
  Interventions: Procedure: control
- IPS group (Active Comparator): patients will receive an ultrasound-guided anterior iliopsoas muscle space (IPS) block
  Interventions: Procedure: IPS
- Supra-iliac QL group (Active Comparator): patients will receive an ultrasound-guided supra-iliac anterior quadratus lumborum (QL) block
  Interventions: Procedure: Supra-iliac QL

INTERVENTIONS:
Procedure: control — patient will be operated under general anesthesia
  Arms: control group
Procedure: IPS — patients will receive ultrasound-guided anterior IPS block with 30 ml of bupivacaine 0.25% followed by general anesthesia.
  Other Names: anterior iliopsoas muscle space block
  Arms: IPS group
Procedure: Supra-iliac QL — patients will receive ultrasound-guided supra-iliac anterior QL block with 30 ml of bupivacaine 0.25% followed by general anesthesia.
  Other Names: supra-iliac anterior quadratus lumborum block
  Arms: Supra-iliac QL group

SUMMARY:
Approximately 1.66 million hip fractures happen in a year worldwide. About 95% of these fractures happen in individuals older than 60 years. Surgical treatment involving THA is considered the best option for patients with hip fractures and those with degenerative changes in the hip joint, especially in the elderly, however, it is associated with moderate to severe postoperative pain.

Pain is one of the main factors limiting ambulation, increasing the risk of thromboembolism by immobility, and causing metabolic changes that affect other systems. Therefore, individualized pain management with the use of appropriate analgesia techniques is of paramount importance. Moreover, early intervention of rehabilitation aiming at a better postoperative recovery may reduce the length of hospital stay and return to daily. Effective pain management is one of the crucial components of enhanced recovery after surgery (ERAS).

Numerous regional anesthetic techniques have been used to provide analgesia following THA, including intrathecal morphine, epidural analgesia, fascia iliaca block, lumber plexus block, sacral plexus block, and local inﬁltration analgesia, however, each of these techniques has specific limitations that prevent them from being the analgesic technique of choice for THA.

Up to investigators' knowledge, there is no study done to compare the supra-iliac approach to the anterior QL block versus the Anterior iliopsoas muscle space block as pre-emptive analgesia in patients undergoing THA under general anesthesia

DETAILED DESCRIPTION:
The acetabulum and the head of the femur combine to produce a traditional ball and socket joint in the hip. The lumbar (L1-L4) and sacral (L4-S4) plexuses both innervate the hip joint, and its sensory innervation is from the femoral (FN), obturator, and sciatic nerves with contribution from the superior gluteal nerve and nerve to quadratus femoris. Cutaneous innervation is by lateral femoral cutaneous (LFCN), subcostal iliohypogastric nerve, and the superior cluneal nerves which predominately arise from the dorsal rami of L1.

The lumbar plexus nerves, including the femoral, obturator, and lateral femoral cutaneous nerves, lie within the psoas major (PM) muscle. These nerves then exit the PM to lie within the iliopsoas compartment, between the iliacus and PM muscles. The sacral plexus is located also in the caudal extension of this anatomical space. The iliacus and psoas muscles are wrapped by the fascia iliaca. The fascia iliaca fuses superiorly with the anterior thoracolumbar fascia (transversalis fascia) that wrapped both the quadratus lumborum (QL) and the psoas muscles.

Total hip arthroplasty (THA) is a common orthopedic surgical procedure that has been successfully utilized to treat hip fractures since 1960 [4] as well, it is considered the treatment of choice for osteoarthritis of the hip joint. Both implants' types cemented and uncemented can provide good fixation, resulting in favorable long-term outcomes [5]. One of the keys to a patient's recovery following THA surgery is effective postoperative pain management. Nowadays, the concept of pain management with multimodal analgesia and regional anesthesia plays a crucial role in postoperative analgesia reducing opioids consumption and decreasing the time to mobilization. Numerous regional anesthetic techniques have been used, including patient-controlled epidural analgesia, intrathecal morphine, fascia iliaca block, lumber plexus block, sacral plexus block, and local inﬁltration analgesia. However, each of these techniques has specific limitations that prevent them from being the analgesic technique of choice for THA.

The ultrasound-guided (QL) block is a regional anesthetic technique that was initially proposed as an analgesic modality for abdominal surgery through many approaches: the lateral QL (QL1) block, the posterior QL (QL2) block, and the anterior QL (transmuscular) block The anterior QL block has been performed at the L3-L4 level also been used in hip surgery case reports.

A supra-iliac approach to the anterior QL block that is performed at a lower level than traditional anterior QL block approaches is considered a new approach discovered by Elsharkawy et al., and they found that a single injection between QL and Psoas muscle at the level of L5, successfully block the lumbar plexus and provide analgesia in patients undergoing total hip arthroplasty.

Anterior iliopsoas muscle space block is a new fascial block technique proposed by Dong et al., where the nerves of the lumbar plexus can be blocked by anterior injection in the iliopsoas space at the level of the anterior superior iliac spine and effectively provide perioperative analgesia for hip surgery.

This study will be designed to evaluate and compare the impact of these two fascial plane blocks for pre-emptive analgesia for patients undergoing total hip arthroplasty under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patient acceptance.
* Age 50-80 years old.
* BMI ≤ 30 kg/m2
* ASA I - III.
* Elective total hip arthroplasty under general anesthesia.

Exclusion Criteria:

* History of allergy to the LA agents used in this study
* Skin lesion at the needle insertion site,
* Those with bleeding disorders, sepsis, liver disease, and psychiatric disorders
* Pre-existing neurological deficit in the lower extremity
* History of chronic pain and taking analgesics
* History of cognitive dysfunction or mental illness

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
changes in Visual analogue scale (VAS)score | measured at 1 hour, 3 hours,6 hours,12hours,18hours, 24 hours postoperatively
  On a scale of 0-10, the patient will learn to quantify postoperative pain where 0= No pain and 10= Maximum worst pain

SECONDARY OUTCOMES:
Total dose of rescue analgesia | in the first 24 hours postoperatively
  once the VAS score will be ≥ 3, rescue analgesia in the form of 1 μg/kg fentanyl will be given and the total dose consumed will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Shereen E Abd Ellatif, MD, Principal Investigator — Faculty of medicine, zagazig university
Locations (1):
- Faculty of medicine, zagazig university, Zagazig, Alsharqia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
planned after the completion of the study and publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: planned after the completion of the study and publication
Access Criteria: contact with principal investigator

REFERENCES:
- [Background] Elsharkawy H, El-Boghdadly K, Barnes TJ, Drake R, Maheshwari K, Soliman LM, Horn JL, Chin KJ. The supra-iliac anterior quadratus lumborum block: a cadaveric study and case series. Can J Anaesth. 2019 Aug;66(8):894-906. doi: 10.1007/s12630-019-01312-z. Epub 2019 Mar 11. PMID 30953311
- [Background] Dong J, Zhang Y, Chen X, Ni W, Yan H, Liu Y, Shi H, Jiang W, Zhao D, Xu T. Ultrasound-guided anterior iliopsoas muscle space block versus posterior lumbar plexus block in hip surgery in the elderly: A randomised controlled trial. Eur J Anaesthesiol. 2021 Apr 1;38(4):366-373. doi: 10.1097/EJA.0000000000001452. PMID 33492871
- [Background] Chalacheewa, T, Termpornlert, S, Sa-Ngasoongsong P, Sangkum, Lisa. Regional Anesthesia for Hip Surgery Patients: Review Article. Journal of the Medical Association of Thailand 2022; 105: 152-9.
- [Background] Dangle J, Kukreja P, Kalagara H. Review of Current Practices of Peripheral Nerve Blocks for Hip Fracture and Surgery. Curr Anesthesiol Rep 2020; 10:259-66.
- [Background] Hockett MM, Hembrador S, Lee A. Continuous Quadratus Lumborum Block for Postoperative Pain in Total Hip Arthroplasty: A Case Report. A A Case Rep. 2016 Sep 15;7(6):129-31. doi: 10.1213/XAA.0000000000000363. PMID 27513972